CLINICAL TRIAL: NCT04307563
Title: Behavioral Health Support for Health Care Providers During COVID 19: A Remote Mindfulness Intervention
Brief Title: Effects of Mindfulness Training on Burnout and Mood in Hospital Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maria Juarez-Reyes, Assistant Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-54792
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Anxiety Depression; Burnout
Keywords: self-compassion; meditation; health personnel
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness group (Other): Participants will attend 6 weekly educational and mindfulness sessions.
  Interventions: Behavioral: Mindfulness session

INTERVENTIONS:
Behavioral: Mindfulness session — 1.5 hour weekly session with health educator

SUMMARY:
The primary aims of the study are to 1) provide a hospital employee population with a mindfulness based stress reduction workshop and 2) evaluate the impact of this clinically validated group mindfulness intervention on burnout in health care employees. Secondary outcomes will be anxiety, depression, quality of life and self compassion.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Employees of Stanford Health Care
* Ability to attend a minimum of 4 out of 6 sessions

Exclusion Criteria:

* Non-English speaking
* Employees with severe medical or psychiatric conditions that prevent them from participating in the group format

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Burnout | Four time points (week 1 and 6 of intervention, and 3 & 6 month post intervention)
  1. Differences in Burnout scale between time points
  The Burnout Scale has been validated by Trockel et al. (2018).It is composed of two subscales (emotional exhaustion containing 4 questions and interpersonal disengagement containing 6 questions.) Both scales are scored on a Likert scale of 0 to 4 ("not at all" to "extremely"). For total Burnout score, the scores of the combined scale (10 total) are averaged. The higher scores indicate higher levels of overall burnout. Individual subscale means will also be computed (with higher scores indicating higher amounts of emotional exhaustion and interpersonal disengagement. Difference in overall burnout measured at four time points (week 1 and 6 of the intervention and 3 & 6 months post intervention) will be reported and compared. The composite scales take approximately 2 minutes to complete.

SECONDARY OUTCOMES:
Change in Anxiety | Four time points (week 1 and 6 of intervention, and 3 & 6 month post intervention)
  1. Differences in GAD-7 between time points.
  The Generalized Anxiety Disorder-7 is a well validated seven-item self-administered questionnaire used to measure anxiety. It has 7 questions with Likert scores ranging from "not at all" (score 0), "several days" (score 1), "more than half the days" (score 2), and "nearly every day (score 3). Scores range from 0 to 21 with higher scores indicating higher levels of anxiety, and a cutoff of or above 10 representing high likelihood of generalized anxiety disorder. Differences in GAD-7 measured at four time points (week 1 and 6 of the intervention and 3 & 6 months post intervention) will be reported and compared. The scale takes approximately 2 minutes.
Change in Depression | Four time points (week 1 and 6 of intervention, and 3 & 6 month post intervention)
  1. Differences in CES-D between time points.
  The Center for Epidemiological Studies - Depression scale is a well validated self-administered questionnaire used to measure depression. The 20 item scale has Likert scores ranging from "rarely or none of the time" (score 0), "some or little of the time" (score 1), "moderate or much of the time" (score 2), and "most or almost all the time" (score 3). Scores range from 0 to 60 with higher scores indicated greater depressive symptoms. A cut off at or above 20 has sensitivity 79% and specificity of 80% for major depression. Difference in CES-D in 2019 measured at four time points (week 1 and 6 of the intervention and 3 & 6 month post intervention) will be reported and compared. The scale takes approximately 5 minutes to complete.
Change in Perceived Health | Four time points (week 1 and 6 of intervention, and 3 & 6 month post intervention)
  1. Differences in GSRH between time points.
  A single item of the Health Related Quality of Life - 4 questionnaire "In general, would you say your health is Excellent (score 1), Very Good (score 2), Good (score 3), Fair (score 4), or Poor (score 5), the general self-rated health (GSRH), is a strong predictor of future health care utilization and mortality. It also has excellent validity. Higher scores of the GSRH are related to higher health care expenditures. Difference in GSRH measured at four time points (week 1 and 6 of the intervention and 3 & 6 month post intervention) will be reported and compared. The scale takes less than 1 minute to complete.
Change in compassion | Four time points (week 1 and 6 of intervention, and 3 & 6 months post intervention)
  1. Differences in compassion scores between time points.
  The 12 item Self-Compassion Scale - Short Form is strongly validated scale to measure self-compassion or "the ability to hold one's feelings of suffering with a sense of warmth, connection and concern". Higher levels of self-compassion are associated with less depression and anxiety. Five-point Likert score are from 1 ("Almost Never") to 5 ("Almost Always"). Total score is computed by reverse scoring negative items of self-judgement, isolation and over-identification (ie 1=5, 2=4, 3=3, 4=2, 5=1) and computing total mean. Difference in Compassion measured at four time points (week 1 and 6 of the intervention, and 3 & 6 month post intervention) will be reported and compared. The scale takes approximately 5-10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Juarez-Reyes, Principal Investigator — Stanford University; Alexandria Blacker, Study Director — Stanford University
Locations (1):
- Stanford Health Care, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazarko D, Cate RA, Azocar F, Kreitzer MJ. The Impact of an Innovative Mindfulness-Based Stress Reduction Program on the Health and Well-Being of Nurses Employed in a Corporate Setting. J Workplace Behav Health. 2013 Apr;28(2):107-133. doi: 10.1080/15555240.2013.779518. PMID 23667348
- [Background] Aiken LH, Clarke SP, Sloane DM, Sochalski J, Silber JH. Hospital nurse staffing and patient mortality, nurse burnout, and job dissatisfaction. JAMA. 2002 Oct 23-30;288(16):1987-93. doi: 10.1001/jama.288.16.1987. PMID 12387650
- [Background] Vollestad J, Nielsen MB, Nielsen GH. Mindfulness- and acceptance-based interventions for anxiety disorders: a systematic review and meta-analysis. Br J Clin Psychol. 2012 Sep;51(3):239-60. doi: 10.1111/j.2044-8260.2011.02024.x. Epub 2011 Sep 9. PMID 22803933
- [Background] Hoge EA, Bui E, Marques L, Metcalf CA, Morris LK, Robinaugh DJ, Worthington JJ, Pollack MH, Simon NM. Randomized controlled trial of mindfulness meditation for generalized anxiety disorder: effects on anxiety and stress reactivity. J Clin Psychiatry. 2013 Aug;74(8):786-92. doi: 10.4088/JCP.12m08083. PMID 23541163
- [Background] DeSalvo KB, Jones TM, Peabody J, McDonald J, Fihn S, Fan V, He J, Muntner P. Health care expenditure prediction with a single item, self-rated health measure. Med Care. 2009 Apr;47(4):440-7. doi: 10.1097/MLR.0b013e318190b716. PMID 19238099
- [Background] Zich JM, Attkisson CC, Greenfield TK. Screening for depression in primary care clinics: the CES-D and the BDI. Int J Psychiatry Med. 1990;20(3):259-77. doi: 10.2190/LYKR-7VHP-YJEM-MKM2. PMID 2265888
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982